CLINICAL TRIAL: NCT00830115
Title: Efficacy of Pantoprazole in Patients Older Than 12 Years With Reflux Associated Sleep Disorders
Brief Title: Pantoprazole 20/40 mg in the Treatment of Symptomatic Reflux Disease With Focus on Sleep Disorders
Acronym: PANDA
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Medical Director, Nycomed Deutschland GmbH
Other Study IDs: P2-9999-010-DE
Record Dates: First submitted 2009-01-13; First posted 2009-01-27 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Sleep Disorders; Non-Erosive Reflux Disease; Gastroesophageal Reflux Disease
Keywords: PPI therapy; Pantoprazole; eGERD (Erosive Gastroesophageal Reflux Disease); NERD (Non-Erosive Reflux Disease)
MeSH Terms: conditions — Sleep Wake Disorders; Non-Erosive Reflux Disease; Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pantoprazole: All patients enrolled
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Observational, non-interventional study (NIS). The physician decided about dosage according to individual needs (20 or 40 mg pantoprazole, once daily).

SUMMARY:
The aim of the study was to evaluate the effect of pantoprazole on sleep disorders in patients with NERD (non-erosive reflux disease) or eGERD (erosive gastroesophageal reflux disease). The prevalence and intensity of the sleep disorders were evaluated by a standardized questionnaire. The study was expected to provide further data on safety and tolerability of pantoprazole.

ELIGIBILITY:
Main inclusion criteria:

* Outpatients with erosive gastro-esophageal reflux disease (eGERD) or non-erosive reflux disease (NERD)

Main exclusion criteria:

* Criteria as defined in the respective Summary of Product Characteristics (Chapter 4.3)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 1045 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bethke, MD, MBA, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (169):
- Germany (169):
  - Nycomed Deutschland GmbH, Aachen
  - Nycomed Deutschland GmbH, Ahrensburg
  - Nycomed Deutschland GmbH, Altenburg
  - Nycomed Deutschland GmbH, Ansbach
  - Nycomed Deutschland GmbH, Aschaffenburg
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Bad Bederkesa
  - Nycomed Deutschland GmbH, Bad Doberan
  - Nycomed Deutschland GmbH, Bad Essen
  - Nycomed Deutschland GmbH, Bad Kissigen
  - Nycomed Deutschland GmbH, Bassum
  - Nycomed Deutschland GmbH, Beckum-Neubeckum
  - Nycomed Deutschland GmbH, Bergkamen
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bietigheim
  - Nycomed Deutschland GmbH, Bitterfeld-Wolfen
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bodenwerder
  - Nycomed Deutschland GmbH, Bovenden
  - Nycomed Deutschland GmbH, Bramsche
  - Nycomed Deutschland GmbH, Brandenburg
  - Nycomed Deutschland GmbH, Bredstedt
  - Nycomed Deutschland GmbH, Bremen
  - Nycomed Deutschland GmbH, Bremerhaven
  - Nycomed Deutschland GmbH, Butzbach
  - Nycomed Deutschland GmbH, Castrop-Rauxel
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Clenze
  - Nycomed Deutschland GmbH, Coburg
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Cölbe
  - Nycomed Deutschland GmbH, Crailsheim
  - Nycomed Deutschland GmbH, Darmstadt
  - Nycomed Deutschland GmbH, Deggendorf
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Dinkelsbühl
  - Nycomed Deutschland GmbH, Dippoldswalde
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Eisenach
  - Nycomed Deutschland GmbH, Ellefeld
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Erlenbach
  - Nycomed Deutschland GmbH, Eschweiler
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Esslingen am Neckar
  - Nycomed Deutschland GmbH, Flensburg
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Freiburg im Breisgau
  - Nycomed Deutschland GmbH, Freising
  - Nycomed Deutschland GmbH, Freudenstadt
  - Nycomed Deutschland GmbH, Fürstenzell
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Gardelegen
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Goch
  - Nycomed Deutschland GmbH, Goslar
  - Nycomed Deutschland GmbH, Greifsfeld
  - Nycomed Deutschland GmbH, Greifswald
  - Nycomed Deutschland GmbH, Grevenbroich
  - Nycomed Deutschland GmbH, Grimmen
  - Nycomed Deutschland GmbH, Großaitingen
  - Nycomed Deutschland GmbH, Güstrow
  - Nycomed Deutschland GmbH, Halberstadt
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Harra
  - Nycomed Deutschland GmbH, Haßfurt
  - Nycomed Deutschland GmbH, Haßloch
  - Nycomed Deutschland GmbH, Hechingen
  - Nycomed Deutschland GmbH, Heide
  - Nycomed Deutschland GmbH, Henstedt-Ulzburg
  - Nycomed Deutschland GmbH, Hildesheim
  - Nycomed Deutschland GmbH, Hof
  - Nycomed Deutschland GmbH, Holzgerlingen
  - Nycomed Deutschland GmbH, Ibbenbueren
  - Nycomed Deutschland GmbH, Johanngeorgenstadt
  - Nycomed Deutschland GmbH, Karlstadt am Main
  - Nycomed Deutschland GmbH, Kassel
  - Nycomed Deutschland GmbH, Kelkheim
  - Nycomed Deutschland GmbH, Kiel
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Kornwestheim
  - Nycomed Deutschland GmbH, L.-E.-Musberg
  - Nycomed Deutschland GmbH, Landstuhl
  - Nycomed Deutschland GmbH, Leer
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Lichtenfels
  - Nycomed Deutschland GmbH, Limburg
  - Nycomed Deutschland GmbH, Lingen
  - Nycomed Deutschland GmbH, Ludwigsfelde
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Ludwigshaven-Oggersheim
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Lüdenscheid
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Marienberg
  - Nycomed Deutschland GmbH, Marl
  - Nycomed Deutschland GmbH, Merseburg
  - Nycomed Deutschland GmbH, Merzig-Schwemlingen
  - Nycomed Deutschland GmbH, Mettlach
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, Möckmühl
  - Nycomed Deutschland GmbH, Mönchnegladbach
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münzenberg
  - Nycomed Deutschland GmbH, Neckargemünd
  - Nycomed Deutschland GmbH, Neu Wulmstorf
  - Nycomed Deutschland GmbH, Neu-Isenburg
  - Nycomed Deutschland GmbH, Neukirchen
  - Nycomed Deutschland GmbH, Neuruppin
  - Nycomed Deutschland GmbH, Neustadt an der Orla
  - Nycomed Deutschland GmbH, Neustadt in Sachsen
  - Nycomed Deutschland GmbH, Nieder-Olm
  - Nycomed Deutschland GmbH, Nordhausen
  - Nycomed Deutschland GmbH, Oberhausen
  - Nycomed Deutschland GmbH, Oberndorf
  - Nycomed Deutschland GmbH, Ochsenfurt
  - Nycomed Deutschland GmbH, Oelsnitz/Erzgeb.
  - Nycomed Deutschland GmbH, Oldenburg
  - Nycomed Deutschland GmbH, Paderborn
  - Nycomed Deutschland GmbH, Papenburg
  - Nycomed Deutschland GmbH, Penig
  - Nycomed Deutschland GmbH, Plauen
  - Nycomed Deutschland GmbH, Plettenberg
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Recklinghausen
  - Nycomed Deutschland GmbH, Regensburg
  - Nycomed Deutschland GmbH, Remscheid
  - Nycomed Deutschland GmbH, Riesa
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Rottach
  - Nycomed Deutschland GmbH, Rottweil
  - Nycomed Deutschland GmbH, Saarbrücken
  - Nycomed Deutschland GmbH, Saarlouis
  - Nycomed Deutschland GmbH, Saint Blasien
  - Nycomed Deutschland GmbH, Salzgitter
  - Nycomed Deutschland GmbH, Schiffweiler
  - Nycomed Deutschland GmbH, Schmalkalden
  - Nycomed Deutschland GmbH, Schwarmstedt
  - Nycomed Deutschland GmbH, Schwäbisch Hall
  - Nycomed Deutschland GmbH, Schwerin
  - Nycomed Deutschland GmbH, Sondeshausen
  - Nycomed Deutschland GmbH, Spaichingen
  - Nycomed Deutschland GmbH, Steinfurt
  - Nycomed Deutschland GmbH, Steißlingen
  - Nycomed Deutschland GmbH, Stockach
  - Nycomed Deutschland GmbH, Strausberg
  - Nycomed Deutschland GmbH, Sundern
  - Nycomed Deutschland GmbH, Tapfheim
  - Nycomed Deutschland GmbH, Varel
  - Nycomed Deutschland GmbH, Waghäusel
  - Nycomed Deutschland GmbH, Wangen
  - Nycomed Deutschland GmbH, Wanzleben
  - Nycomed Deutschland GmbH, Weißenburg
  - Nycomed Deutschland GmbH, Weißenfels
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Willich
  - Nycomed Deutschland GmbH, Wismar
  - Nycomed Deutschland GmbH, Wittenberg
  - Nycomed Deutschland GmbH, Zell
  - Nycomed Deutschland GmbH, Zerbst
  - Nycomed Deutschland GmbH, Zweibrücken
  - Nycomed Deutschland GmbH, Zwickau

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients were evaluated, missing values were not imputed.
Period: Overall Study
Arm/Group | Pantoprazole
Started | 1045
Completed | 1042
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Improvement/recovery | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1045
Age Continuous [Mean (Standard Deviation); unit: years] — The measured value is related to the number of 1041 subjects (= valid cases). This number differs from the overall number of baseline participants due to missing data for 4 subjects.
  years | 52.9 (15.39)
Sex/Gender, Customized [Number; unit: participants]
  Female | 480
  Male | 563
  Missing data | 2
Alcohol use [Number; unit: participants]
  Daily | 173
  Not daily | 862
  Missing data | 10
Diagnosis: reflux disease [Number; unit: participants]
  NERD (Non-Erosive Reflux Disease) | 393
  eGERD (Erosive Gastro-Esophageal Reflux Disease) | 649
  Missing Data | 3
Drug abuse [Number; unit: participants]
  Drug abuse | 14
  No drug abuse | 1016
  Missing data | 15
Nicotine use [Number; unit: participants]
  Smoker | 342
  Non-smoker | 685
  Missing data | 18

OUTCOME MEASURES:

1. Primary Outcome: Patient's Assessment of Stanford Sleepiness Scale for the Last 24 Hours (Diaries)
Description: Assessment on a scale from 1=Feeling active, vital, alert, or wide awake to 7=No longer fighting sleep, sleep onset soon, having dream-like thoughts
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 869
  * Day 1 = 868
  * Day 2 = 867
  * Day 3 = 864
  * Day 4 = 863
  * Day 5 = 859
  * Day 6 = 862
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Pantoprazole: All patients with valid value at least at day 0
Arm/Group | Pantoprazole
Number analyzed (Participants) | 869
Units on a scale
  Day 0 | 2.94 (1.58)
  Day 1 | 2.62 (1.41)
  Day 2 | 2.28 (1.23)
  Day 3 | 2.03 (1.12)
  Day 4 | 1.86 (1.06)
  Day 5 | 1.74 (1.02)
  Day 6 | 1.67 (1.01)

2. Primary Outcome: Patient's Assessment of Sleep Disturbances for the Last 24 Hours (Diaries)
Description: Assessment on a scale: Severity from 1=Not impaired to 10=Severely impaired
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 846
  * Day 1 = 841
  * Day 2 = 828
  * Day 3 = 817
  * Day 4 = 800
  * Day 5 = 791
  * Day 6 = 790
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 846
Units on a scale
  Day 0 | 3.65 (2.39)
  Day 1 | 3.07 (2.11)
  Day 2 | 2.53 (1.84)
  Day 3 | 2.21 (1.65)
  Day 4 | 2.00 (1.54)
  Day 5 | 1.78 (1.42)
  Day 6 | 1.68 (1.34)

3. Primary Outcome: Physician's Assessment of Sleep Disturbances
Description: Assessment on a scale: 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 7 days
Population: Patients included and treated with valid data at first and last visit (without imputation of missing values), intention to treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Pantoprazole: All patients with valid values at first and last visit
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1011
Units on a scale
  Start of therapy | 2.03 (0.94)
  End of study | 1.26 (0.54)

4. Secondary Outcome: Patient's Assessment of General Well-being for the Last 24 Hours (Diaries)
Description: Assessment on a scale: Severity from 1=Excellent to 10=Extremely bad
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 908
  * Day 1 = 906
  * Day 2 = 890
  * Day 3 = 876
  * Day 4 = 861
  * Day 5 = 842
  * Day 6 = 834
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 908
Units on a scale
  Day 0 | 5.23 (2.26)
  Day 1 | 4.45 (2.14)
  Day 2 | 3.62 (1.96)
  Day 3 | 2.98 (1.77)
  Day 4 | 2.53 (1.63)
  Day 5 | 2.26 (1.61)
  Day 6 | 2.05 (1.52)

5. Secondary Outcome: Patient's Assessment of Acid Complaints for the Last 24 Hours (Diaries)
Description: Assessment on a scale: Severity from 1=Not impaired to 10=Severely impaired
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 903
  * Day 1 = 891
  * Day 2 = 877
  * Day 3 = 843
  * Day 4 = 823
  * Day 5 = 791
  * Day 6 = 781
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 903
Units on a scale
  Day 0 | 5.75 (2.35)
  Day 1 | 4.37 (2.25)
  Day 2 | 3.22 (2.01)
  Day 3 | 2.53 (1.65)
  Day 4 | 2.05 (1.42)
  Day 5 | 1.70 (1.16)
  Day 6 | 1.49 (1.08)

6. Secondary Outcome: Patient's Assessment of Upper-abdominal/Stomach Complaints for the Last 24 Hours (Diaries)
Description: Assessment on a scale: Severity from 1=Not impaired to 10=Severely impaired
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 887
  * Day 1 = 867
  * Day 2 = 846
  * Day 3 = 823
  * Day 4 = 801
  * Day 5 = 784
  * Day 6 = 773
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 887
Units on a scale
  Day 0 | 4.47 (2.51)
  Day 1 | 3.56 (2.20)
  Day 2 | 2.72 (1.90)
  Day 3 | 2.25 (1.59)
  Day 4 | 1.89 (1.40)
  Day 5 | 1.67 (1.32)
  Day 6 | 1.49 (1.16)

7. Secondary Outcome: Patient's Assessment of Lower Abdominal/Digestive Complaints for the Last 24 Hours (Diaries)
Description: Assessment on a scale: Severity from 1=Not impaired to 10=Severely impaired
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 798
  * Day 1 = 782
  * Day 2 = 769
  * Day 3 = 759
  * Day 4 = 752
  * Day 5 = 739
  * Day 6 = 738
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 798
Units on a scale
  Day 0 | 2.64 (2.12)
  Day 1 | 2.31 (1.84)
  Day 2 | 1.94 (1.53)
  Day 3 | 1.76 (1.35)
  Day 4 | 1.62 (1.26)
  Day 5 | 1.50 (1.23)
  Day 6 | 1.42 (1.12)

8. Secondary Outcome: Patient's Assessment of Nausea for the Last 24 Hours (Diaries)
Description: Assessment on a scale: Severity from 1=Not impaired to 10=Severely impaired
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 809
  * Day 1 = 798
  * Day 2 = 776
  * Day 3 = 761
  * Day 4 = 743
  * Day 5 = 738
  * Day 6 = 732
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 809
Units on a scale
  Day 0 | 3.22 (2.46)
  Day 1 | 2.52 (2.03)
  Day 2 | 2.07 (1.68)
  Day 3 | 1.78 (1.41)
  Day 4 | 1.60 (1.30)
  Day 5 | 1.42 (1.11)
  Day 6 | 1.30 (1.03)

9. Secondary Outcome: Physician's Assessment of Heartburn
Description: Assessment on a scale: 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 7 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1022
Units on a scale
  Start of therapy | 3.05 (0.75)
  End of study | 1.33 (0.56)

10. Secondary Outcome: Physician's Assessment of Acid Eructation
Description: Assessment on a scale: 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 7 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1019
Units on a scale
  Start of therapy | 2.77 (0.83)
  End of study | 1.25 (0.50)

11. Secondary Outcome: Physician's Assessment of Painful Swallowing
Description: Assessment on a scale: 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 7 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1017
Units on a scale
  Start of therapy | 1.76 (0.87)
  End of study | 1.07 (0.30)

12. Secondary Outcome: Assessment of the Efficacy of Pantoprazole at Final Visit
Description: Assessment on a scale: 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 7 days
Population: Patients included and treated with at least one application of pantoprazole (without imputation of missing values), intention to treat
Measure: Number; unit: Participants
Groups:
- Pantoprazole: Patients included and treated with at least one application of pantoprazole
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1045
Participants
  Excellent | 719
  Good | 246
  Satisfactory | 30
  Not satisfactory | 11
  Missing data | 39

13. Secondary Outcome: Assessment of the Tolerability of Pantoprazole at Final Visit
Description: Assessment on a scale: 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 7 days
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1045
Participants
  Excellent | 847
  Good | 150
  Satisfactory | 7
  Not satisfactory | 4
  Missing data | 37

ADVERSE EVENTS:
Time Frame: First until last intake (planned 7 days)
Arm/Group | Pantoprazole
Serious Adverse Events (participants affected / at risk) | 0/1045
Other Adverse Events (participants affected / at risk) | 4/1045
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole (N=1045)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No